CLINICAL TRIAL: NCT02241876
Title: EVALUATION OF THE USE OF N-ACETYLCYSTEINE ATTENUATING CISPLATIN-INDUCED TOXICITIES BY OXIDATIVE STRESS IN HEAD AND NECK CANCER PATIENTS
Brief Title: THE USE OF N-ACETYLCYSTEINE ATTENUATING CISPLATIN-INDUCED TOXICITIES BY OXIDATIVE STRESS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Patricia Moriel, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NAC+Cisplatin2014
Record Dates: First submitted 2014-09-05; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): The patients will be treated with placebo as follows: 15 mL (0 mg of drug), once a day, during 7 days in each cycle (2 days before chemotherapy with cisplatin, on the day of chemotherapy and more 4 days after chemotherapy).
- N-Acetylcysteine (Experimental): The patients will be treated with n-acetylcysteine as follows: 15 mL (600mg of drug), once a day, during 7 days in each cycle (2 days before chemotherapy with cisplatin, on the day of chemotherapy and more 4 days after chemotherapy).
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine
  Arms: N-Acetylcysteine

SUMMARY:
Head and neck cancer corresponds to tumors located in the upper aerodigestive tract, such as the oral cavity, pharynx and larynx. The most effective treatment consists of high dose of cisplatin chemotherapy and radiotherapy, however, their use is limited due to toxicities caused mainly by oxidative stress. The objective of this study will be evaluate the use of n-acetylcysteine attenuating cisplatin-induced toxicities by oxidative stress in head and neck cancer patients. This is a randomized double-blind placebo-controlled clinical trial with consecutive sampling that will be conducted at Oncology Department of Clinic Hospital / University of Campinas (UNICAMP). Head and neck cancer patients who will begin cisplatin antineoplastic treatment (80-100mg/m2 on days 1, 22 and 43) and concurrent radiotherapy will be included in this research. They will be studied in 2 groups (n-acetylcysteine and placebo). All patients will be evaluated in relation to cisplatin induced hematologic and gastrointestinal disorders, nephrotoxicity, ototoxicity, and hepatotoxicity; plasmatic and cellular oxidative stress; quality of life; and pharmacoeconomic evaluation. Results will be statistically analysed using Chi-square, Fisher, Mann-Whitney, and ANOVA for repeated measures tests (p<0.05.)

ELIGIBILITY:
Inclusion Criteria:

* head and neck cancer
* anticancer treatment - cisplatin (80 to 100 mg/m²) plus radiotherapy
* patients without previous treatment of head and neck cancer (surgery, chemotherapy and radiotherapy)

Exclusion Criteria:

* severe psychiatric diseases
* impossibility of verbal communication
* without caregivers or companions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Hematologic, Nephro, and Hepato Toxicity - Degree of toxicity by Common Toxicity Criteria for Adverse Effects (CTCAE - version 4.0) | 120 hours
  Hematologic - anemia, leukopenia, neutropenia, lymphopenia, thrombocytopenia; Nephrotoxicity - increase of serum creatinine level and reduction of creatinine clearance; Hepatotoxicity - increase of AST, ALT, ALP, GGT, Total Bilirubin levels.
  The time frame is 120 hours post-dose and 20 days post-dose (each cycle of Chemotherapy)
Gastrointestinal Toxicity - Degree of toxicity by CTCAE (version 4.0) | 1 day
  Nausea, Vomiting and Diarrhea The time frame is on day 1 and up to 120 hours post-dose (each cycle)
audiometric testing | 1 day
  audiometric testing for identification of ototoxic hearing loss. The time frame is prior to day 1 and 30 days after treatment completion
Nephrotoxicity | 1 day
  The nephrotoxicity will be evaluated by EDTA-51Cr. The time frame are prior to day 1 and 30 days after treatment completion

SECONDARY OUTCOMES:
Quality of Life | 21 days
  Quality of Life by EORTC-QLQ- 30 and EORTC-QLQ-H&N35 questionnaires The time frame are Day, 1, 22, 43, and 21 days after treatment completion
Cellular and plasma oxidative stress biomarkers | 1 day
  Time frame are Before day 1; 120 hours post-dose and 20 days post-dose (each cycle of chemotherapy)
Effectiveness of anticancer therapy | 1 day
  The effectiveness of anticancer therapy will be analyzed by Computed Tomography of the head and neck. The time frame are prior to day 1 and 30 days after treatment completion

CONTACTS AND LOCATIONS:
Locations (1):
- State University of Campinas - UNICAMP, Hospital das Clinicas, Campinas, São Paulo, Brazil